CLINICAL TRIAL: NCT07019857
Title: Impact of Thymectomy on Immune Response in Infants 12 Months After Cardiac Surgery: a Single-centre Prospective Study
Brief Title: Impact of Thymectomy on Immunity in Infants After Cardiac Surgery
Acronym: THYMIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC24_0411
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Defects; Thymectomy; Immunological Deficiency Syndrome
Keywords: Thymectomy; Cardiac Surgery; Infant; Immunity; Lymphocytes; TRECs; Vaccination; Infection
MeSH Terms: conditions — Heart Defects, Congenital; Immunologic Deficiency Syndromes; Infections

STUDY DESIGN:
Intervention Model Description: three groups according to type of surgery (complete thymectomy, partial thymectomy, control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complete Thymectomy Group (Experimental): Infants undergoing cardiac surgery with cardiopulmonary bypass (CPB), during which a complete thymectomy is performed for surgical access to the heart and great vessels. The extent of thymus resection is determined by the cardiac surgeon intraoperatively, based on anatomical considerations
  Interventions: Diagnostic Test: Blood sample collection at surgery time and 12 months later
- Partial Thymectomy Group (Experimental): Infants undergoing cardiac surgery with CPB, during which a partial thymectomy is performed, with an effort to preserve thymic tissue when anatomically feasible.
  Interventions: Diagnostic Test: Blood sample collection at surgery time and 12 months later
- Control Group (No Thymectomy (Active Comparator): Infants undergoing:
  * Cardiac surgery by thoracotomy without thymectomy (e.g., for aortic coarctation) or
  * Non-cardiac surgery (e.g., digestive procedures) with complete preservation of the thymus.
  These patients serve as immunological reference controls
  Interventions: Diagnostic Test: Blood sample collection at surgery time and 12 months later

INTERVENTIONS:
Diagnostic Test: Blood sample collection at surgery time and 12 months later — each participant undergoes a blood test 1) at surgery time and 2) 12 months after surgery. These 5mL samples include:
  * Blood cell count
  * TREC dosage
  * Complete Lymphocytes immunophenotyping
  * Immunoglobulin dosage

SUMMARY:
Heart surgery in infants typically involves complete removal of the thymus gland to improve access to the heart. However, the thymus plays a key role in developing the immune system in early childhood, especially in the production and maturation of T lymphocytes, which help the body defend itself against infections.

The THYMIC study tests the hypothesis that partial removal of the thymus (partial thymectomy) during heart surgery may better preserve the child's immune function compared to total removal (complete thymectomy). The goal is to determine whether this conservative surgical approach could reduce the risk of immune system impairment and infections in the months following surgery.

This is a prospective, interventional, single-center study conducted at CHU de Nantes, involving 3 groups of infants:

* One group undergoing heart surgery with complete thymectomy;
* One group undergoing heart surgery with partial thymectomy;
* One control group undergoing heart or non-heart surgery without thymus removal. All infants enrolled will have two blood tests: one taken during their surgery and one taken one year later. These blood tests will quantify immune cells (T, B, NK cells), levels of antibodies, and vaccine responses. Parents will also be asked to fill out a questionnaire to record any infections their child experiences during the year after surgery.

By comparing the immune responses and infection rates among the groups, the researchers hope to better understand the long-term effects of thymectomy in infants. The results could support future recommendations to preserve part of the thymus when possible during heart surgery.

Participation in the study does not change the medical or surgical care of the child. The decision to perform a partial or complete thymectomy is made by the surgeon based on the child's anatomy. The additional blood samples are small in volume and follow current safety regulations.

DETAILED DESCRIPTION:
The THYMIC study is a prospective, single-center, interventional clinical trial conducted at the University Hospital of Nantes (CHU de Nantes), France. It aims to evaluate the medium-term immunological impact of thymectomy (total versus partial) in infants undergoing cardiac surgery requiring cardiopulmonary bypass (CPB) before the age of 6 months.

Background and Rationale During most pediatric cardiac surgeries, the thymus is completely removed to allow better access to the heart and great vessels. However, the thymus plays a critical role in T-cell development during infancy, contributing to immune system maturation. Prior studies suggest that complete thymectomy in early life may result in persistent alterations in T-cell immunity and increased susceptibility to infections. Yet, the comparative impact of partial versus complete thymectomy on immune function remains poorly studied.

Partial thymectomy is technically feasible in selected cases depending on the anatomy, and could offer a balance between surgical access and immune preservation. The THYMIC study tests the hypothesis that partial thymectomy is associated with less impairment of cellular immunity at 12 months postoperatively and could therefore become the preferred surgical approach in appropriate cases.Study Design

This is a non-randomized, controlled study including 70 infants:

• 50 infants undergoing cardiac surgery with CPB and either partial or complete thymectomy (surgical decision made

The THYMIC study is a prospective, single-center, interventional clinical trial conducted at the University Hospital of Nantes (CHU de Nantes), France. It aims to evaluate the medium-term immunological impact of thymectomy (total versus partial) in infants undergoing cardiac surgery requiring cardiopulmonary bypass (CPB) before the age of 6 months.

Background and Rationale During most pediatric cardiac surgeries, the thymus is completely removed to allow better access to the heart and great vessels. However, the thymus plays a critical role in T-cell development during infancy, contributing to immune system maturation. Prior studies suggest that complete thymectomy in early life may result in persistent alterations in T-cell immunity and increased susceptibility to infections. Yet, the comparative impact of partial versus complete thymectomy on immune function remains poorly studied.

Partial thymectomy is technically feasible in selected cases depending on the anatomy, and could offer a balance between surgical access and immune preservation. The THYMIC study tests the hypothesis that partial thymectomy is associated with less impairment of cellular immunity at 12 months postoperatively and could therefore become the preferred surgical approach in appropriate cases.

Study Design

This is a non-randomized, controlled study including 70 infants:

* 50 infants undergoing cardiac surgery with CPB and either partial or complete thymectomy (surgical decision made intraoperatively),
* 10 infants undergoing cardiac surgery via thoracotomy without thymectomy (control group A),
* 10 infants undergoing non-cardiac surgery (e.g., digestive surgery) without thymectomy (control group B).

The study involves two blood draws:

* Baseline (preoperative): performed at anesthesia induction via central catheter (5 mL), including blood cell counts, lymphocyte immunophenotyping, immunoglobulin levels, and TRECs (if Guthrie test not already available).
* Follow-up (12 months postoperative): peripheral blood draw (5 mL), with repeated immunophenotyping, immunoglobulin levels, and post-vaccine serologies (e.g., diphtheria, tetanus, pneumococcus).

Parents are given a standardized infection monitoring questionnaire at hospital discharge, to be completed with their pediatrician or other care providers over the 12-month follow-up. A phone call is scheduled at 6 months to reinforce compliance. At 12 months, families return for the second blood draw and review of the infection questionnaire. An additional consultation is conducted 15 days later to provide results and arrange follow-up if needed.

Primary Objective To compare cellular immune profiles at 12 months between infants with partial versus complete thymectomy. Key markers include absolute counts of lymphocytes and subsets, and T-cell receptor excision circles (TRECs).

Secondary Objectives

To compare:

* Humoral immunity markers (B-cell subsets, immunoglobulin levels, vaccine responses),
* Clinical outcomes such as the number, type, and severity of infections (e.g., hospitalization, ICU admission, antibiotic use) between groups.

Methodology Notes Due to the impossibility of preoperative randomization (surgical decision on thymectomy extent depends on intraoperative anatomy), this is a non-randomized study with group allocation based on surgical findings.

All data are pseudonymized and collected in an electronic case report form (eCRF). Immunological assays are processed via the CHU's certified laboratories (CIMNA platform and hematology department).

Ethical Considerations and Risk-Benefit Assessment The study poses minimal risk. Blood samples are within safe volume limits for infants, and pain is minimized using anesthetic cream and inhaled analgesia (EMLA, MEOPA). Thymectomy extent is based solely on clinical indication and does not depend on study participation. Families benefit from enhanced immunological monitoring, which could identify and help manage acquired immune deficiencies.

Significance This study may provide critical data to support a shift toward more conservative surgical practices regarding thymus preservation in early cardiac surgery, with the potential to reduce long-term immunological sequelae in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* - Children aged between 0 and 6 months;
* Born at a gestational age > 37 weeks' gestation;
* With an indication for cardiac surgery under CEC at Nantes University Hospital;
* Cardiopediatric follow-up planned at Nantes University Hospital;
* Written agreement signed by legal guardians to participate in the study.

For the control groups:

* Control group A (cardiac surgery without thymectomy):

  * Children aged between 0 and 6 months of age;
  * Born at a gestational age > 37 SA;
  * Indicated for thoracotomy cardiac surgery at Nantes University Hospital;
  * Cardiopediatric follow-up planned at Nantes University Hospital;
  * Written agreement signed by legal guardians to participate in the study.
* Control group B (non-cardiac surgery)

  * Children aged between 0 and 6 months;
  * Born at a gestational age > 37 SA;
  * Indicated for non-cardiac surgery (ENT or visceral surgery at Nantes University Hospital);
  * Planned follow-up surgery at Nantes University Hospital;
  * Written agreement signed by legal guardians to participate in the study.

Exclusion Criteria :

* Gestational age < 37 SA;
* With a history of cardiac surgery under ECG;
* And/or with heart disease requiring further surgery within 12 months of the 1st surgery (e.g. pulmonary cerclage, systemic pulmonary anastomosis).
* And/or a history of partial or complete thymectomy;
* Receiving long-term immunosuppressive treatment;
* Post-operative follow-up planned in a hospital other than Nantes University Hospital, or moving house planned during the follow-up period;
* parental refusal.

Exclusion Criteria:

* - Gestational age < 37 SA;
* With a history of cardiac surgery under ECG;
* And/or with heart disease requiring further surgery within 12 months of the 1st surgery (e.g. pulmonary cerclage, systemic pulmonary anastomosis).
* And/or a history of partial or complete thymectomy;
* Receiving long-term immunosuppressive treatment;
* Post-operative follow-up planned in a hospital other than Nantes University Hospital, or moving house planned during the follow-up period;
* parental refusal.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
T-Lymphocyte response | 12 months after surgery
  biological endpoint with absolute quantification of LyTs, LyT subpopulations and TRECs.

SECONDARY OUTCOMES:
Humoral response | 12 months after surgery
  absolute quantification of LyB, weighted immunoglobulin assays and post-vaccination serologies
Clinical impact | 12 months after surgery
  the number of infectious episodes, their severity as assessed by the need for hospitalisation, the number of days spent in intensive care, the number of days on antibiotics, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Chenouard, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No